CLINICAL TRIAL: NCT03057964
Title: The Effect of Combined Treatment of PDL and Fractional Photothermolysis on the Cosmetic Appearance of Postsurgical Scars
Brief Title: PDL and Fractional Photothermolysis for Postsurgical Scars
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology-Head and Neck Surgery, and Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00204024
Record Dates: First submitted 2017-02-09; First posted 2017-02-20 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Scar
MeSH Terms: conditions — Cicatrix | interventions — Lasers, Dye

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- PDL (Pulsed Dye Laser) and Fractional Photothermolysis (Experimental)
  Interventions: Device: PDL (Pulsed Dye Laser); Device: Fractional Photothermolysis Laser
- Control (No Intervention)

INTERVENTIONS:
Device: PDL (Pulsed Dye Laser) — For those in the experimental group, at each treatment visit, the subject's scar will be treated with PDL followed by fractional photothermolysis.
  Other Names: Pulsed Dye Laser
  Arms: PDL (Pulsed Dye Laser) and Fractional Photothermolysis
Device: Fractional Photothermolysis Laser — For those in the experimental group, at each treatment visit, the subject's scar will be treated with PDL followed by fractional photothermolysis.
  Other Names: Fraxel Laser
  Arms: PDL (Pulsed Dye Laser) and Fractional Photothermolysis

SUMMARY:
This is a two part study to evaluate the efficacy of early combined PDL (pulsed dye laser) and fractional photothermolysis in the cosmetic improvement of post surgical scars.All subjects will be offered at the time of the dermatologic procedure, an option to treat the post surgical scars with early combined PDL and fractional photothermolysis.

Part A is a non-randomized study design and subjects will have the choice of whether or not they will receive treatment. In part B, subjects will be randomized in a 2:1 treatment vs. control design.

The experimental group will have a total of 6 visits: 1 standard of care suture removal visit, 3 treatment visits and 2 follow up visits. The control group will have 3 visits: 1 standard of care suture removal visit and 2 follow up visits.

Subjects currently living in the Chicago metropolitan area and meet inclusion/exclusion criteria will be considered for enrollment.

This study is a pilot study designed to determine feasibility of this procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 18 years old
2. Fitzpatrick skin types I-VI
3. Subjects are in good health as judged by the investigator.
4. Subjects who have received dermatologic surgery procedure of the trunk or extremities closed with complex primary closure with subcuticular running suture removed at 2-3 weeks.
5. Subjects applying topical retinoids, must discontinue one week prior to treatment.
6. Subjects who are willing and have the ability to understand and provide informed consent for participation in the study and are able to communicate with the investigator.

Exclusion Criteria:

1. History of recurrent facial or labial herpes simplex infection
2. Subjects applying topical retinoids, must discontinue one week prior to treatment.
3. Subjects with a history of hypertrophic scars or keloids
4. Pregnant or breast feeding
5. Uncooperative patients or patients with neurological disorders who are incapable of following directions or who are predictably unwilling to return for follow-up examinations.
6. Subjects who are unable to understand the protocol or give informed consent.
7. Subjects who in the opinion of the investigator are likely to have exaggerated scarring with laser treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in score of Patient and Observer Scar Assessment Scale (POSAS) | Baseline and 6 Months
  The POSAS is a series of questions about the scar with a scale from 1 to 10 with 1 as "not at all" or "normal skin" and 10 as "very much so" or "very different".

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kang BY, Ibrahim SA, Weil A, Reynolds KA, Johnson T, Wilson S, Lee MH, Kim JYS, Dirr MA, Poon E, Alam M. Treatment of Surgical Scars With Combination Pulsed Dye and Fractional Nonablative Laser: A Randomized Controlled Trial. Ann Surg. 2022 Dec 1;276(6):975-980. doi: 10.1097/SLA.0000000000005377. Epub 2022 Jan 25. PMID 35081564